CLINICAL TRIAL: NCT03496363
Title: Evaluation of Thyroid Function in Children With Congenital Heart Disease
Brief Title: Hypothyroidism With Congenital Heart Disease (CHD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa M Atteya, Principal investigator, Assiut University
Other Study IDs: CHD
Record Dates: First submitted 2018-03-10; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Hypothyroidism; CHD
Keywords: Children
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHD with Hypothyroidism
  Interventions: Diagnostic Test: TSH , T4

INTERVENTIONS:
Diagnostic Test: TSH , T4 — Thyroid stimulating hormone

SUMMARY:
Congenital hypothyroidism is one of the most preventable causes of neurocognitive impairment because early treatment is possible in neonates. The thyroid hormone is important for normal growth and development in infancy. After introducing national screening test using capillary thyroid stimulating hormone level, the incidence of untreated congenital hypothyroidism has significantly decreased.

According to the Italian Registry of Congenital Hypothyroidism, congenital heart disease is the most frequent disease condition associated with congenital hypothyroidism.

Congenital heart disease is also reported to be a risk factor for non-autoimmune hypothyroidism in children. In addition, intravenous iodine contrast media is frequently used for diagnostic imaging and therapeutic intervention in congenital heart disease patients. Excess iodine exposed by iodine contrast media may disturb thyroid function in adult and pediatric population. However, there is no generally accepted guideline for screening thyroid dysfunction in congenital heart disease infants.

An increased prevalence of thyroid disease, particularly sub-clinical hypothyroidism, has been reported in Down Syndrome. In children with Down Syndrome, a possible concomitant sub-clinical hypothyroidism-related impairment of cardiac function or structure may worsen their clinical condition and can ultimately affect their life expectancy.

DETAILED DESCRIPTION:
Aim of the work :

The aim of the work is to assess the thyroid function in children with congenital heart disease.

Inclusion criteria :

Patients with congenital heart diseases from birth (full term) to 3 years.

Exclusion criteria :

Patients with cardiac disease other than congenital heart disease. Preterm infants. Patients with other non cardiac congenital anomalies. Other endocrinal or central nervous system dysfunction. Maternal history of thyroid disease or antithyroid management.

Methods :

The study will be conducted in the Cardiology or Neonatology Units , Children's University Hospital, Faculty of Medicine, Assiut University on 50 patients both males and females.

All children will be evaluated by thoroughly history taken. Full general (including the anthropometric measures) and cardiac examinations will be done.

The patients will be conducted to investigations as:

Thyroid function tests. Electrocardiograph. X-ray chest and heart. Echocardiography.

Ethical considerations:

1. Risk benefit assessment, All patients will not be subjected to risk of any kind during this study.
2. Confidentiality, All patient's data will be confidential and stored in a secure location.
3. Informed consent, An informed consent will be taken from all patients and included.
4. Other ethical consideration, The research will be conducted only by scientifically qualified and trained personnel

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital heart diseases from birth (full term) to 3 years

Exclusion Criteria:

* Patients with cardiac disease other than congenital heart disease
* Preterm infants
* Patients with other non cardiac congenital anomalies
* Other endocrinal or CNS dysfunction
* Maternal history of thyroid disease or antithyroid management

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
EVALUATE THYROID FUNCTION IN PATIENTS WITH CONGENITAL HEART DISEASE | May 2018 - May 2020
  The study include evaluation of Thyroid function in patients with congenital heart disease coming to cardiology unit - pediatric hospital - Assiut University by measuring TSH and T4 level and detect percentage of hypothyroidism in patients with congenital heart disease.

SECONDARY OUTCOMES:
Detect the percentage of patients with congenital heart disease and have no thyroid problems | May 2018 - May 2020
  If TSH and T4 level in patients with congenital heart disease is in normal value , then detect the percentage of patients with congenital heart disease and have no thyroid problems.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gruters A, Krude H. Detection and treatment of congenital hypothyroidism. Nat Rev Endocrinol. 2011 Oct 18;8(2):104-13. doi: 10.1038/nrendo.2011.160. PMID 22009163
- [Background] Rastogi MV, LaFranchi SH. Congenital hypothyroidism. Orphanet J Rare Dis. 2010 Jun 10;5:17. doi: 10.1186/1750-1172-5-17. PMID 20537182
- [Background] Oerbeck B, Sundet K, Kase BF, Heyerdahl S. Congenital hypothyroidism: influence of disease severity and L-thyroxine treatment on intellectual, motor, and school-associated outcomes in young adults. Pediatrics. 2003 Oct;112(4):923-30. doi: 10.1542/peds.112.4.923. PMID 14523187
- [Background] Leger J, Larroque B, Norton J; Association Francaise pour le Depistage et la Prevetion des Handicaps de l'Enfant. Influence of severity of congenital hypothyroidism and adequacy of treatment on school achievement in young adolescents: a population-based cohort study. Acta Paediatr. 2001 Nov;90(11):1249-56. doi: 10.1080/080352501317130272. PMID 11808894
- [Background] American Academy of Pediatrics; Rose SR; Section on Endocrinology and Committee on Genetics, American Thyroid Association; Brown RS; Public Health Committee, Lawson Wilkins Pediatric Endocrine Society; Foley T, Kaplowitz PB, Kaye CI, Sundararajan S, Varma SK. Update of newborn screening and therapy for congenital hypothyroidism. Pediatrics. 2006 Jun;117(6):2290-303. doi: 10.1542/peds.2006-0915. PMID 16740880
- [Background] Olivieri A, Stazi MA, Mastroiacovo P, Fazzini C, Medda E, Spagnolo A, De Angelis S, Grandolfo ME, Taruscio D, Cordeddu V, Sorcini M; Study Group for Congenital Hypothyroidism. A population-based study on the frequency of additional congenital malformations in infants with congenital hypothyroidism: data from the Italian Registry for Congenital Hypothyroidism (1991-1998). J Clin Endocrinol Metab. 2002 Feb;87(2):557-62. doi: 10.1210/jcem.87.2.8235. PMID 11836285
- [Background] Passeri E, Frigerio M, De Filippis T, Valaperta R, Capelli P, Costa E, Fugazzola L, Marelli F, Porazzi P, Arcidiacono C, Carminati M, Ambrosi B, Persani L, Corbetta S. Increased risk for non-autoimmune hypothyroidism in young patients with congenital heart defects. J Clin Endocrinol Metab. 2011 Jul;96(7):E1115-9. doi: 10.1210/jc.2011-0057. Epub 2011 Apr 27. PMID 21525159
- [Background] Barr ML, Chiu HK, Li N, Yeh MW, Rhee CM, Casillas J, Iskander PJ, Leung AM. Thyroid Dysfunction in Children Exposed to Iodinated Contrast Media. J Clin Endocrinol Metab. 2016 Jun;101(6):2366-70. doi: 10.1210/jc.2016-1330. Epub 2016 Mar 28. PMID 27018967
- [Background] Ahmet A, Lawson ML, Babyn P, Tricco AC. Hypothyroidism in neonates post-iodinated contrast media: a systematic review. Acta Paediatr. 2009 Oct;98(10):1568-74. doi: 10.1111/j.1651-2227.2009.01412.x. Epub 2009 Jul 3. PMID 19575766
- [Background] Lee SY, Rhee CM, Leung AM, Braverman LE, Brent GA, Pearce EN. A review: Radiographic iodinated contrast media-induced thyroid dysfunction. J Clin Endocrinol Metab. 2015 Feb;100(2):376-83. doi: 10.1210/jc.2014-3292. Epub 2014 Nov 6. PMID 25375985
- [Background] Toscano E, Pacileo G, Limongelli G, Verrengia M, Di Mita O, Di Maio S, Salerno M, Del Giudice E, Caniello B, Calabro R, Andria G. Subclinical hypothyroidism and Down's syndrome; studies on myocardial structure and function. Arch Dis Child. 2003 Nov;88(11):1005-8. doi: 10.1136/adc.88.11.1005. PMID 14612370